CLINICAL TRIAL: NCT04521790
Title: Role of Endomyocardial Biopsy and Aetiology-based Treatment in Patients With Inflammatory Heart Disease in Arrhythmic and Non-arrhythmic Clinical Presentations: an Integrated Approach for the Optimal Diagnostic and Therapeutic Management
Acronym: MYOCAR
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Peretto, MD, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: MYOCAR
Record Dates: First submitted 2020-07-01; First posted 2020-08-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myocarditis; Ventricular Arrythmia; Inflammatory Cardiomyopathy; Genetic Predisposition; Autoimmunity; Arrhythmia; Cardiomyopathies; Immunosuppression; Catheter Ablation
Keywords: Myocarditis; Ventricular arrhythmias; Arrhythmias; Arrhythmogenic inflammatory cardiomyopathy; Endomyocardial biopsy; Cardiac magnetic resonance; Ablation; Positron emission tomography; Cardiac imaging; Electroanatomical mapping; Immunosuppressive therapy; Arrhythmic risk stratification; Genetic predisposition; Environment; Implantable cardioverter defibrillator; Implantable loop recorder; Multicenter
MeSH Terms: conditions — Myocarditis; Genetic Predisposition to Disease; Autoimmune Diseases; Arrhythmias, Cardiac; Cardiomyopathies | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Undefined a-priori. Will be considered in clinically-indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arrhythmic (A): Arrhythmic Group. To oversimplify, specific subgroups of patients will be considered.
  1. Group 1: major ventricular arrhythmias (haemodynamically unstable VT, hu-VT; ventricular fibrillation, VF).
  2. Group 2: other ventricular arrhythmias (high-burden premature ventricular complexes = hb-PVC; nonsustained VT = NSVT; haemodynamically stable VT = hs-VT).
  3. Group 3: bradyarrhythmias (2nd type II or 3rd degree atrioventricular block = advanced AVB; critical sinus pauses = SND).
  4. Group 4: supraventricular arrhythmias (atrial fibrillation = AF; atrial flutter = AFlu; atrial tachycardia = AT).
  Interventions: Other: support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation
- Nonarrhythmic (NA): Nonarrhythmic Group. To oversimplify, specific subgroups of patients will be considered.
  1. Heart failure presentation (and subtypes)
  2. Chest pain presentation (and subtypes)
  3. Asymptomatic presentation/screening (and subtypes)
  Interventions: Other: support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation
- Subgroups: For specific study aims, different patient subgroups will be compared. The main groups are hereby reported:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…).
  C. Infectious vs. autoimmune vs. toxic myocarditis. D. Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment.
  E. Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis.
  F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease.
  G. Myocarditis vs. peri-myocarditis/myo-pericarditis. H. Other subgroups.
  Interventions: Other: support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation

INTERVENTIONS:
Other: support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation — Treatment will be patient-tailored, integrating international guidelines recommendation and the experience of the center where enrollment takes place.

SUMMARY:
Myocarditis is a complex inflammatory disease, usually occurring secondary to viral infections, autoimmune processes or toxic agents. Clinical presentations are multiple, including chest-pain, heart failure and a broad spectrum of arrhythmias. In turn, outcome is largely unpredictable, ranging from mild self-limiting disease, to chronic stage and progressive evolution towards dilated cardiomyopathy, to rapid adverse outcome in fulminant forms. Subsequently, myocarditis is often underdiagnosed and undertreated, and optimal diagnostic and therapeutic strategies are still to be defined. This study, both retrospective and prospective, originally single-center and subsequently upgraded to multicenter, aims at answering multiple questions about myocarditis, with special attention to its arrhythmic manifestations.

1. Optimal diagnostic workflow is still to be defined. In fact, although endomyocardial biopsy (EMB) is still the diagnostic gold standard, especially for aetiology identification, it is an invasive technique. Furthermore, it may lack sensitivity because of sampling errors. By converse, modern imaging techniques - cardiac magnetic resonance (CMR) in particular - have been proposed as alternative or complementary diagnostic tool in inflammatory heart disease. Other noninvasive diagnostic techniques, like delayed-enhanced CT (DECT) scan or position emission tomography (PET) scan, are under investigation.
2. Biomarkers to identify myocarditis aetiology, predisposition, prognosis and response to treatment are still to be defined.
3. Arrhythmic myocarditis is largely underdiagnosed and uninvestigated. Importantly, myocarditis presenting with arrhythmias requires specific diagnostic, prognostic and therapeutic considerations. At the group leader hospital, which is an international referral center for ventricular arrhythmias management and ablation, a relevant number of patients with unexplained arrhythmias had myocarditis as underlying aetiology. The experience of a dedicated third-level center is going to be shared with other centers, to considerably improve knowledge and management of arrhythmic myocarditis.
4. The role of CMR, as well as alternative noninvasive imaging techniques, in defining myocarditis healing is a relevant issue. In particular, optimal timing for follow-up diagnostic reassessment is still to be defined, in patients with myocarditis at different inflammatory stages, either with or without aetiology-dependent treatment.
5. Uniformly-designed studies are lacking, to compare myocarditis among different patient subgroups, differing by variables like: clinical presentations, myocarditis stage, associated cardiac or extra-cardiac diseases, aetiology-based treatment, associated arrhythmic manifestations, diagnostic workup, and devices or ablation treatment.

DETAILED DESCRIPTION:
This study, previously designed as a single-center experience, is multicenter, observational and both retrospective and prospective.

Retrospective phase includes all clinical data occurring before the index event (hospitalization or clinically suspected myocarditis) and myocarditis diagnosis. Prospective phase includes all data following index event and myocarditis diagnosis.

This study has multiple aims.

1. To compare EMB with noninvasive diagnostic techniques (CMR, DECT, PET scan, either alone or in association).
2. To assess the role of blood biomarkers for identification of aetiology, predisposition, prognosis, response to treatment, inflammatory activity, clinical presentation.
3. To describe myocarditis presenting with arrhythmias, with special focus on ventricular arrhythmias at different myocarditis stages and in different clinical contexts. To validate and generalize the leader hospital model for optimal diagnostic and therapeutical management of arrhythmias in myocarditis patients (given the role of the leader hospital as an international referral center for arrhythmias ablation and management).
4. To evaluate the timing needed for myocarditis healing in different patients subgroups, as assessed by noninvasive imaging techniques (CMR, DECT, PET scan), either alone or in association.
5. To compare patients subgroups of myocarditis, in terms of epidemiology, aetiology, prognosis, and diagnostic-therapeutical strategies. Among the others, the main study subgroups will be:

A. Arrhythmic vs. non-arrhythmic myocarditis. B. Arrhythmic myocarditis subgroups. C. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…).

D. Infectious vs. autoimmune vs. toxic myocarditis. E. Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment.

F. Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis.

G. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease.

H. Myocarditis vs. peri-myocarditis/myo-pericarditis. I. Other analyses.

Any adult patient with clinically suspected myocarditis, of any clinical presentation and any degree of severity, will be considered as suitable for study enrollment.

Patients will undergo diagnostic and therapeutical strategies considered as clinically indicated in a patient-tailored manner, as suggested by international guidelines recommendations and best local clinical practice. Patients will be free of either accepting or refusing any diagnostic or therapeutical proposal. Whenever accepted, data will be simply collected and analyzed.

Based on clinical presentation, patients will be divided into two groups, arrhythmic (group A) and non-arrhythmic (group NA, including any other clinical presentation).

Independently of A/NA groups, all patients will undergo optimal diagnostic and therapeutic strategies, as summarized in panel A. In parallel, special diagnostic and therapeutical strategies will be performed in patients with arrhythmic presentation or evidence of arrhythmias, as shown in panel B. Proposed flowcharts (Panels A and B) represent only an approximate algorithm. Exceptions can be made in single cases, based on clinical indications.

Panel A - Diagnostic and therapeutical workup in all patients. Independently of groups (A/NA), all patients will undergo optimal diagnostic and therapeutical workup, guided by updated scientific evidence merged with the clinical experience of the center.

Baseline diagnostic workup will include: complete blood exams, 12-leads ECG, continuous telemetric monitoring, transthoracic doppler echocardiogram, coronary artery imaging (coronary angiography or CT scan). Any other clinically relevant diagnostic test will be collected.

In life-threatening presentations (cardiogenic shock or malignant arrhythmias), support treatment by optimal medical therapy, inotropic or mechanical circulatory support, and acute-phase arrhythmia management (including cardioversion, defibrillation, or temporary pacing) will be performed, as indicated, before completing diagnostic workup.

Final diagnosis of myocarditis will include, whenever applicable:

A. For stable patients: 1) a second-level imaging technique (CMR as first choice; and/or DECT, PET, or multiple/fusion imaging techniques, based on clinical indications); followed by: 2) EMB, whenever clinically indicated. Blood exams for aetiology screening will be personalized upon clinical indications.

B. For unstable patients: EMB only, as recommended. Blood exams for aetiology screening will be personalized upon clinical indications.

Diagnostic criteria for myocarditis, as assessed by any diagnostic technique, will be defined based on international scientific evidence and will be constantly updated. Similar considerations apply to myocarditis staging and aetiology definition. Whenever not available at local institutions, diagnostic exams can be performed and analyzed at external centers.

All patients with myocarditis (or any alternative final diagnosis), will undergo standard cardiological optimal medical treatment (COMT), as indicated. By converse, aetiology-dependent treatment will be performed only in patients with a final diagnosis of any active (acute, fulminant, chronic active) myocarditis of defined aetiology (EMB-proved). Multidisciplinary assessment, including infective disease specialists (in viral/infective myocarditis), immunologists (in non-infective/autoimmune myocarditis) or any other specialist as needed, will be used to identify indications to treatment, drug choice (either approved or with a justified unapproved indication), treatment duration and safety profile, aiming at the best patients' interest. Toxic myocarditis will be treated accordingly, by evaluating the opportunity of withdrawing pathogenic noxa.

This protocol will not interfere with local best clinical practice. Patients with non-active myocarditis (previous or healed) or with non-myocarditis, will undergo "standard FU" (see below). Patients with active myocarditis will undergo "intensive FU" (see below).

Independently of FU modalities, diagnostic reassessment will be considered in the presence of at least one of the following instability criteria: a) new unexplained cardiac symptoms (dyspnoea, chest pain, syncope, palpitation); b) new unexplained increase in troponin or natriuretic peptides; c) new imaging abnormal signs; d) new unexplained clinically relevant arrhythmias. Diagnostic reassessment will include second-level imaging and/or EMB, as shown above. Subsequent therapeutical workup will be in line with the above explanations. In stable patients or undergone myocarditis healing, exercise stress test will be obtained, whenever possible.

Panel B - Diagnostic and therapeutical workup of patients with arrhythmias In parallel with (and independently of) Panel A content, patients with arrhythmias (group A) will undergo specific diagnostic and therapeutical management for arrhythmias, as a result of the integration between international guidelines recommendations and the experience of an international referral center for arrhythmia management and ablation.

To oversimplify, 4 groups of patients will be considered.

1. Group 1: major ventricular arrhythmias, including haemodynamically unstable VT (hu-VT) and ventricular fibrillation (VF).

   After electrical stabilization and support treatment (panel A), indication to secondary prevention ICD implant will be multiparametric and patient-tailored. In patients with active myocarditis, subcutaneous ICD (S-ICD) or wearable CD (WCD) will be considered. Antiarrhythmic drugs will be considered in all Group 1 patients. In addition, all Group 1 patients will undergo COMT and aetiology-dependent treatment whenever applicable (panel A). Ablation of ventricular arrhythmias will be considered in patients with severe arrhythmic presentation, or symptomatic, or refractory to optimal medical treatment. Electrophysiological study (EPS) may be used in selected cases. A cardiac resynchronization therapy with defibrillator function (CRT-D) will replace ICD whenever indicated.
2. Group 2: other ventricular arrhythmias, including high-burden (hb) premature ventricular complexes (PVC); nonsustained VT (NSVT); haemodynamically stable VT (hs-VT).

   Whenever clinically indicated, Group 2 patients will undergo invasive EPS (or in alternative noninvasive programmed ventricular stimulation in ICD carriers) to stratify arrhythmic risk. Patients with positive EPS will undergo ICD (or S-ICD/WCD) as in Group 1. Patients with negative EPS, as well as Group 2 cases not undergoing EPS, will undergo watchful waiting strategy (always with an intensive FU) with or without loop recorder implant: in these cases, ICD (or S-ICD/WCD) will be implanted only following documentation of relevant VA in FU. In addition, all Group 2 patients will undergo antiarrhythmic treatment, COMT and aetiology-dependent treatment whenever applicable (panel A). In symptomatic or drug-refractory cases, ablation of ventricular arrhythmias will be considered. A CRT-D will replace ICD whenever indicated.
3. Group 3: bradyarrhythmias, including advanced (2nd type II or 3rd degree) atrioventricular block (AVB); critical sinus pauses from sinus node disease (SND).

   After electrical stabilization and support treatment (panel A), including the use of temporary pacemaker as a bridge-to-decision, patients will undergo watchful waiting strategy or definitive device implant. Instead of a pacemaker (PM), ICD will be considered in the presence of high-risk criteria for ventricular tachyarrhythmias, including: a) overlap with Group 1 presentation; b) overlap with Group 2 presentation, especially in the presence of positive EPS; c) other indications for primary prevention ICD implant (severe systolic dysfunction); d) signs of increased tachyarrhythmic risk (scar signs); e) patients with special aetiologies leading to an increased tachyarrhythmic risk (i.e: cardiac sarcoid, giant cell myocarditis, Chagas disease, overlapping genetic syndromes). In addition, all Group 3 patients will undergo COMT and aetiology-dependent treatment whenever applicable (panel A). A CRT-D or a CRT-P will replace ICD or PM, respectively, whenever indicated.
4. Group 4: supraventricular arrhythmias, including atrial fibrillation (AF); atrial flutter (AFlu); atrial tachycardia (AT).

   Following acute-phase rate control (RaC), stable rhythm control (RyC) strategy will be considered as the therapeutical target, together with appropriate anticoagulation, as needed. Normal sinus rhythm will be obtained through either electrical or pharmacological cardioversion. In patients with unsuccessful attempts of sinus rhythm conversion, optimal treatment of active myocarditis will be considered as a primary target. Following myocarditis healing, in the presence of persistent arrhythmias, patients will be considered for RyC via electrical or pharmacological cardioversion. Transcatheter ablation will be an option for patients with drug-symptomatic, recurrent or refractory arrhythmias. Permanent RaC strategy will be considered only in non responders. Widespread use of implantable loop recorders will apply, as clinically indicated. In addition, all Group 4 patients will undergo COMT and aetiology-dependent treatment whenever applicable (panel A).

   Aims in detail. Aim 1 Comparison between EMB and second level imaging findings (N=1000)

   Primary:

   Diagnostic concordance

   Secondary:

   Inflammatory activity (presence; type; quantification) Fibrosis (presence; type; quantification) Coronary microvascular disease Comparison between EMB sampling site and abnormal substrate localization at imaging (including substrate-guided EMB or alternative biopsy techniques) Role of EMB guided by electroanatomical map Diagnostic performance of DECT and/or PET, especially when CMR is contraindicated Comparison between CMR/DECT findings and PET scan (including fusion imaging) or advanced imaging techniques including strain analysis at echocardiogram Comparison between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) Comparison among different diagnostic techniques (EMB, CMR/DECT, PET) in terms of safety and diagnostic accuracy Evaluation of differential diagnosis with other cardias diseases, and particularly with arrhythmogenic cardiomyopathy of any localization (left, right, biventricular, to identify updated diagnostic criteria) Comparison between information provided by all the techniques above, and data from electroanatomical mapping (EAM) Other analyses

   Aim 2 Evaluation of blood exams and biomarkers (N=1000)

   Primary:

   Identification of diagnostic biomarkers Identification of aetiology biomarkers

   Secondary:

   Cardiac and inflammatory biomarkers evaluation in different myocarditis subtypes Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) Comparison between local and systemic/peripheral inflammation Correlations with EMB and second-level imaging (CMR, DECT, PET…) findings Identification of genetic factors with any role in predisposition, prognosis, response to treatment, or any other correlation, either in the presence or in the absence of underlying cardiomyopathy or autoimmune/inflammatory disease Identification of prognostic biomarkers Identification of biomarkers associated with treatment response Evaluation of any tissue/organ damage or associated comorbidities Study of cardiac autoantibodies Study of any cell, tissue, genetic or circulating biomarker Correlations with clinical presentations Other analyses

   Aim 3 Validation of optimal management of arrhythmic myocarditis (N=1000)

   Primary:

   Evaluation of effects on major endpoints

   Secondary:

   Evaluation of effects on minor endpoints Role of electrophysiological study in risk stratification Role of loop recorders in arrhythmia monitoring Role of transcatheter ablation (any technique) on arrhythmic outcomes Identification of optimal timing for any electrophysiological/device procedure Role of pharmacological antiarrhythmic treatment Role of aetiology-specific treatment on arrhythmic outcomes Identification of criteria for device implants (PM, ICD, S-ICD, CRT-D…) in myocarditis patients Validation of therapeutic strategies and their optimal timing in patients with supraventricular arrhythmias, bradyarrhythmias, or ventricular arrhythmias Correlation between arrhythmia type/features with any other diagnostic exam performed at baseline or during FU (mainly EMB, CMR/DECT/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell biomarkers) Indications and timing for device (ICD, CRT-D) implant in primary prevention, based on multiparametric risk assessment, and in relation to different general and aetiology-dependent treatments Other analyses

   Aim 4 Evaluation of healing timing in myocarditis (N=500) Primary Any degree of recovery by 3, 6, 9, 12 and > 12 months Secondary Comparison of healing times in treated vs. untreated patients Correlations between healing times and clinical presentation types Correlations between healing times and any biomarker Correlations between healing times and any outcomes Validation of exercise stress test role after myocarditis healing Evaluation of PET scan or other diagnostic techniques as alternatives to CMR in special populations Other analyses

   Aim 5 Subgroup analyses (N=500, hugely variable in each subanalysis) A vs. NA groups; A myocarditis subgroups; NA myocarditis subgroups (including fulminant); Infective vs. autoimmune vs. toxic forms; Treated by aetiology-driven therapy vs. standard cardiological treatment; Different myocarditis stages and differential diagnoses; Isolated vs. in the context o a systemic disease or genetic disease; Myocarditis vs. perimyocarditis/ myopericarditis Primary Differences in major outcomes Secondary Differences in minor outcomes Differences in any biomarker Differences in any diagnostic exam Differences in aetiology Differences in predisposition Differences in inflammatory activity Differences in pericardial involvement Differences in systemic involvement Differences in arrhythmias types and features Differences in clinical presentation Differences in treatment response, including novel treatments Validation of local aetiology/pathophysiology-dependent treatments Validation of biomarkers and imaging techniques in monitoring response to treatment Identification of optimal follow-up timeline Other analyses

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age ≥ 18 years.
* Clinically suspected myocarditis.
* Enrollment performed by one of the participating Centers.

Exclusion Criteria:

* Absence of written informed consent.
* Age < 18 years (paediatric population).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will enroll adult patients (age ≥ 18 y), of any gender or ethnic group, evaulated for clinically suspected myocarditis. Patients can be enrolled from any medical environment or department, including inpatients, outpatients, and patients transferred from other hospitals. The same inclusion criteria of the original single-center protocol will apply to the entire multicenter study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major cardiac events | By 12-month follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Occurrence of major cardiac events | By 24-month follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Occurrence of major cardiac events | By 3-year follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Occurrence of major cardiac events | By 5-year follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Occurrence of major cardiac events | By 7-year follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Occurrence of major cardiac events | By 10-year follow-up
  death; cardiac death; malignant ventricular arrhythmias ( = VT, VF, appropriate ICD therapy); heart transplantation; end-stage heart failure
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | At baseline assessment
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 6-month follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 12-month follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 24-month follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 3-year follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 5-year follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) between EMB and second level imaging findings - Primary | By 10-year follow-up
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Comparison of troponin values in patients with different aetiologies | At baseline assessment
  Measurement of troponin blood concentration (ng/l) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Description of troponin values changes during follow-up | By 10-year follow-up
  Measurement of troponin blood concentration (ng/l) during follow-up, and description of its relative variation compared to baseline assessment.
Comparison of creatine-phosphokinase values in patients with different aetiologies | At baseline assessment
  Measurement of creatine-phosphokinase (U/l) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Description of creatine-phosphokinase values changes during follow-up | By 10-year follow-up
  Measurement of creatine-phosphokinase (U/l) during follow-up, and description of its relative variation compared to baseline assessment.
Comparison of natriuretic peptides values in patients with different aetiologies | At baseline assessment
  Measurement of natriuretic peptides (pg/ml) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Description of natriuretic peptides values changes during follow-up | By 10-year follow-up
  Measurement of natriuretic peptides (pg/ml) during follow-up, and description of its relative variation compared to baseline assessment.
Comparison of C-reactive protein values in patients with different aetiologies | At baseline assessment
  Measurement of C-reactive protein (mg/l) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Description of C-reactive protein values changes during follow-up | By 10-year follow-up
  Measurement of C-reactive protein (mg/l) during follow-up, and description of its relative variation compared to baseline assessment.
Comparison of erythrocyte sedimentation rate values in patients with different aetiologies | At baseline assessment
  Measurement of erythrocyte sedimentation rate (mm/h) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Description of erythrocyte sedimentation rate values changes during follow-up | By 10-year follow-up
  Measurement of erythrocyte sedimentation rate (mm/h) during follow-up, and description of its relative variation compared to baseline assessment.
Comparison of procalcitonin values in patients with different aetiologies | At baseline assessment
  Measurement of procalcitonin (mcg/ml) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of procalcitonin values in patients with different aetiologies | By 10-year follow-up
  Measurement of procalcitonin (mcg/ml) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of serum uric acid values in patients with different aetiologies | At baseline assessment
  Measurement of serum uric acid (mg/dl) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of serum uric acid values in patients with different aetiologies | By 10-year follow-up
  Measurement of serum uric acid (mg/dl) and comparison of values found in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of leukocyte values in patients with different aetiologies | At baseline assessment
  Measurement of leukocytes (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of leukocyte values in patients with different aetiologies | By 10-year follow-up
  Measurement of leukocytes (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of hemoglobin values in patients with different aetiologies | At baseline assessment
  Measurement of hemoglobin (g/dl) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of hemoglobin values in patients with different aetiologies | By 10-year follow-up
  Measurement of hemoglobin (g/dl) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of platelet values in patients with different aetiologies | At baseline assessment
  Measurement of platelets (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of platelet values in patients with different aetiologies | By 10-year follow-up
  Measurement of platelets (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of thyroid function in patients with different aetiologies | At baseline assessment
  Measurement of thyroid stimulating hormone (mU/ml; total and fractions) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of thyroid function in patients with different aetiologies | By 10-year follow-up
  Measurement of thyroid stimulating hormone (mU/ml; total and fractions) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of organ damage in patients with different aetiologies | At baseline assessment
  Measurement of organ damage by application of the Sequential Organ Failure Assessment (SOFA) score in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Comparison of organ damage in patients with different aetiologies | By 10-year follow-up
  Measurement of organ damage by application of the Sequential Organ Failure Assessment (SOFA) score in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of autoimmunity screening | At baseline assessment
  Measurement of circulating autoantibodies (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of autoimmunity screening | By 10-year follow-up
  Measurement of circulating autoantibodies (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of infectious screening | At baseline assessment
  Measurement of viral antibodies (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of infectious screening | By 10-year follow-up
  Measurement of viral antibodies (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of toxicology screening | At baseline assessment
  Measurement of toxic urynalisis (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of toxicology screening | By 10-year follow-up
  Measurement of toxic urynalisis (U/ml) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of genetic test screening | At baseline assessment
  Reporting the results of next generation sequencing analysis (mutation type) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Reporting the results of genetic test screening | By 10-year follow-up
  Reporting the results of next generation sequencing analysis (mutation type) in patients with different aetiologies (viral; autoimmune; toxic; non-myocarditis).
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 10-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 12-month follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 24-month follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 3-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 5-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Validation of optimal management of arrhythmic myocarditis by comparing the occurrence of major cardiac events in patients undergoing different therapeutic strategies - Primary | By 7-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Evaluation of healing timing in myocarditis - Primary | By 1-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 3-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 6-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 9-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 12-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 18-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 24-month follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 3-year follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 5-year follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 7-year follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Evaluation of healing timing in myocarditis - Primary | By 10-year follow-up
  Any degree of recovery through analysis of CMR, other second level imaging, echocardiogram, cardiac and inflammatory biomarkers, symptoms, arrhythmia burden, and exercise tolerance.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | At baseline assessment
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 12-month follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 24-month follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 3-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 5-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 7-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of the incidence of major cardiac events in different patient subgroups - Primary | By 10-year follow-up
  Evaluation of the occurrence of major cardiac events (death; cardiac death; malignant ventricular arrhythmias= VT, VF, appropriate ICD therapy; heart transplantation; end-stage heart failure) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.

SECONDARY OUTCOMES:
Occurrence of minor arrhythmic events | At baseline assessment and through study completion (up to 10 years)
  NSVT; PVC burden; supraventricular arrhythmias; bradyarrhythmias
Any modification in imaging parameters | At baseline assessment and through study completion (up to 10 years)
  Structural or functional myocardial abnormalities at echocardiogram or second level imaging (any chamber dilation, systolic or diastolic dysfunction, including strain analysis, pericardial, vascular or valvular involvement, any other detectable abnormalities; qualitative and quantitative evaluation); signal abnormalities detectable by advanced imaging techniques (Lake Louise criteria and T-mapping techniques at CMR; any qualitative or quantitative imaging abnormality detectable by CMR, DECT or PET scan, or other imaging techniques, alone or in association).
Any modification in clinical parameters | By 10-year follow-up
  Signs and symptoms related to cardiac or multisystemic disease, as assessed by dedicated questionnaires.
Any modification in New York Heart Association class | By 10-year follow-up
  Change in New York Heart Association class (range I-IV; significant change for improvement by at least one class).
Any modification in exercise peak heart rate | By 10-year follow-up
  Reporting changes in exercise peak heart rate (beats per minute) by any cardiac or cardiopulmonary stress test, by comparing follow-up results with baseline performance
Any modification in exercise peak systolic blood pressure | By 10-year follow-up
  Reporting changes in exercise peak systolic blood pressure (mmHg) by any cardiac or cardiopulmonary stress test, by comparing follow-up results with baseline performance
Any modification in exercise walking distance | By 10-year follow-up
  Reporting changes in exercise walking distance (meters) by any cardiac or cardiopulmonary stress test, by comparing follow-up results with baseline performance
Any modification in exercise oxygen consumption | By 10-year follow-up
  Reporting changes in exercise oxygen consumption (l/min) by any cardiac or cardiopulmonary stress test, by comparing follow-up results with baseline performance
Any modification in exercise-induced arrhythmias | By 10-year follow-up
  Reporting changes in exercise-induced arrhythmias (type) by any cardiac or cardiopulmonary stress test, by comparing follow-up results with baseline performance
Identification of the prevalence of associated diseases | By 10-year follow-up
  Identification of any comorbidity associated with myocarditis (qualitative description)
Any modification in arrhythmia burden | By 10-year follow-up
  Change in daily and monthly arrhythmia burden quantification, as compared to baseline assessment
Any modification in arrhythmia morphology | By 10-year follow-up
  Change in 12-lead ECG morphology (QRS axis) of arrhythmias, as compared to baseline assessment
Any modification in arrhythmia regularity | By 10-year follow-up
  Change in arrhythmia cycle length regularity, as compared to baseline
Any modification in arrhythmia tolerance | By 10-year follow-up
  Change in arrhythmia hemodynamic tolerance (presence or absence of syncope), as compared to baseline assessment
Prevalence of coronary circulation abnormalities | By 10-year follow-up
  Reporting the prevalence of any anatomical or functional abnormality found at: coronary angiography; CT scan; histology; provocative stress tests, nuclear medicine techniques
Prevalence of electrophysiological study | By 10-year follow-up
  Reporting prevalence of electrophysiological study in the population, including indication and timing.
Results of electrophysiological study | By 10-year follow-up
  Reporting the results of electrophysiological study (inducibility of ventricular tachycardia or fibrillation), including the association with occurrence of arrhythmias (ventricular tachycardia, ventricular fibrillation, appropriate ICD therapy) during follow-up.
Prevalence of ventricular arrhythmia ablation | By 10-year follow-up
  Reporting prevalence of ventricular arrhythmia ablation in the population, including indication and timing.
Results of ventricular arrhythmia ablation | By 10-year follow-up
  Reporting the results of ventricular arrhythmia ablation (inducibility of ventricular tachycardia or fibrillation at the end of the procedure), including the association with occurrence of arrhythmias (ventricular tachycardia, ventricular fibrillation, appropriate ICD therapy) during follow-up.
Prevalence of supraventricular arrhythmia ablation | By 10-year follow-up
  Reporting prevalence of supraventricular arrhythmia ablation (atrial fibrillation, atrial flutter, atrial tachycardia) in the population, including indication and timing.
Results of supraventricular arrhythmia ablation | By 10-year follow-up
  Reporting the results of supraventricular arrhythmia ablation by assessing the occurrence of supraventricular arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia) during follow-up.
Prevalence of cardiac device implants | By 10-year follow-up
  Reporting prevalence of cardiac device implants (pacemakers, ICD, CRT-P, CRT-D, WCD, S-ICD, implantable loop recorders) in the population, including indication and timing.
Comparison of arrhythmia detection by continuous vs. non-continuous monitoring | By 10-year follow-up
  Assessment of the occurrence of arrhythmias detected by continuous arrhythmia monitoring (pacemakers, ICD, CRT-P, CRT-D, WCD, S-ICD, implantable loop recorders) as compared to those detected by non-continuous arrhythmia monitoring (Holter ECG).
Assessment of the withdrawal timing of non-permanent cardiac devices | By 10-year follow-up
  Reporting the time of witrhdrawal of non-permanent cardiac devices (WCD, S-ICD, loop recorders).
Prevalence of CT scan | By 10-year follow-up
  Reporting prevalence of CT scan in the population, including indication and timing.
Results of CT scan | By 10-year follow-up
  Reporting the results of CT scan (number of positive results; both in absolute, and as compared to the other imaging techniques)
Prevalence of PET scan | By 10-year follow-up
  Reporting prevalence of PET scan in the population, including indication, type and timing.
Results of PET scan | By 10-year follow-up
  Reporting the results of PET scan (number of positive results; both in absolute, and as compared to the other imaging techniques)
Prevalence of electroanatomical mapping | By 10-year follow-up
  Reporting prevalence of electroanatomical mapping in the population, including indication and timing.
Results of electroanatomical mapping | By 10-year follow-up
  Reporting the results of electroanatomical mapping (number of positive results; both in absolute, and as compared to the other imaging techniques)
Prevalence of stress tests | By 10-year follow-up
  Reporting prevalence of stress tests, including indication, type (ECG; echocardiogram; scintigraphy; CMR; 6-minute walking test; cardiac rehabilitation programs; cardiopulmonary stress test) and timing.
Results of stress tests - ECG | By 10-year follow-up
  Reporting the results of stress tests (prevalence of ST segment modification) in the population, including the association with major outcomes (malignant ventricular arrhythmias; heart failure requiring intravenous diuretics, hospitalization, or heart transplantation).
Results of stress tests - wall motion abnormalities | By 10-year follow-up
  Reporting the results of stress tests (prevalence of wall motion abnromalities by either echocardiogram, scintigraphy or CMR) in the population, including the association with major outcomes (malignant ventricular arrhythmias; heart failure requiring intravenous diuretics, hospitalization, or heart transplantation).
Results of stress tests - coronary flow reserve | By 10-year follow-up
  Reporting the results of stress tests (prevalence of reduced coronary flow reserve, as assessed by either scintigraphy, CMR, or PET scan) in the population, including the association with major outcomes (malignant ventricular arrhythmias; heart failure requiring intravenous diuretics, hospitalization, or heart transplantation).
Myocarditis recurrences | At baseline assessment (including past medical history) and through study completion (up to 10 years)
  Reporting of any myocarditis recurrences (either clinically-suspected, biomarker-proven, CMR or second level imaging-proven, or EMB-proven); comparison with first myocarditis episode; investigation of underlying aetiology.
Response to treatment - systolic function | At baseline assessment and through study completion (up to 10 years)
  Comparison of any change in left ventricular ejection fraction (LVEF) in patients undergoing different treatment strategy:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Response to treatment - malignant ventricular arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Comparison of any change in the incidence of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy) in patients undergoing different treatment strategy:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Prognostic risk stratification - malignant ventricular arrhythmias | Through study completion (up to 10 years)
  Identification of independent predictors of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy) during follow-up in the population, as assessed by either univariable or multivariable risk stratification models.
Prognostic risk stratification - heart failure | Through study completion (up to 10 years)
  Identification of independent predictors of heart failure (= hospitalization for acute heart failure, heart transplantation, left ventricular ejection fraction below 35%) during follow-up in the population, as assessed by either univariable or multivariable risk stratification models.
Prognostic risk stratification - cardiac death | Through study completion (up to 10 years)
  Identification of independent predictors of cardiac death during follow-up in the population, as assessed by either univariable or multivariable risk stratification models.
Description of multidisciplinary workup models | At baseline assessment and through study completion (up to 10 years)
  Description of types and number of physicians from different medical specializations involved in the management of myocarditis patients.
Prognostic impact of multidisciplinary workup models | At baseline assessment and through study completion (up to 10 years)
  Comparison of outcomes (cardiac death, heart failure, malignant ventricular arrhythmias) between patients managed by single vs. multiple physicians.
Comparison between EMB and second level imaging findings in detecting myocardial inflammation | At baseline assessment and through study completion (up to 10 years)
  Reporting myocardial inflammation (presence; type; quantification) in EMB vs. second level imaging techniques
Comparison between EMB and second level imaging findings in detecting myocardial fibrosis | At baseline assessment and through study completion (up to 10 years)
  Reporting myocardial fibrosis (presence; type; quantification) in EMB vs. second level imaging techniques
Comparison between EMB and second level imaging findings in detecting coronary microvascular disease | At baseline assessment and through study completion (up to 10 years)
  Reporting coronary microvascular disease (presence; type) in EMB vs. second level imaging techniques
Comparison between EMB sampling site and abnormal substrate localization at imaging | At baseline assessment and through study completion (up to 10 years)
  Descriprion of EMB sampling site in relation to the localization of abnormal substrate as assessed by second level imaging techniques
Comparison between substrate-guided vs. standard EMB sampling. Substrate defined by any second level imaging technique (CMR, PET, DECT, electroanatomical mapping). EMB sampling performed at any cardiac site. | At baseline assessment and through study completion (up to 10 years)
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Comparison between different second level imaging findings | At baseline assessment and through study completion (up to 10 years)
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value. Comparison of substrate abnormalities (localization; pattern; extension; distribution) as found by different second level imaging techniques, including CMR, DECT, PET, electroanatomical mapping, and echocardiogram (including fusion imaging). Scar definition, characterization and composition.Texture analysis.Other analyses.
Associations between arrhythmia morphology and substrate localization | At baseline assessment and through study completion (up to 10 years)
  Identification of association (sensitivity, specificity, positive predictive value, negative predictive value) between arrhythmia morphology pattern (right superior; right inferior; left superior; left inferios - as assessed by 12-lead ECG) and substrate localization (anterior; septal; lateral; inferior - as defined by any second level imaging technique including CMR, PET, DECT, electroanatomical mapping).
Associations between arrhythmia morphology and inflammatory stage | At baseline assessment and through study completion (up to 10 years)
  Identification of association (sensitivity, specificity, positive predictive value, negative predictive value) between arrhythmia mophology (monomorphic vs. polymorphic, as assessed by 12-lead ECG) and inflammatory stage (active vs. nonactive, as assessed by any technique including EMB, CMR, PET, DECT, electroanatomical mapping, troponin)
Associations between arrhythmia regularity and inflammatory stage | At baseline assessment and through study completion (up to 10 years)
  Identification of association (sensitivity, specificity, positive predictive value, negative predictive value) between arrhythmia regularity (regular vs. irregular, as assessed by 12-lead ECG) and inflammatory stage (active vs. nonactive, as assessed by any technique including EMB, CMR, PET, DECT, electroanatomical mapping, troponin)
Prevalence of adverse effects associated with EMB | At baseline assessment and through study completion (up to 10 years)
  Reporting the prevalence of adverse effects (death; pericardial effusion; vascular complications) associated with EMB.
Prevalence of adverse effects associated with immunosuppressive therapy | At baseline assessment and through study completion (up to 10 years)
  Reporting the prevalence of adverse effects (death; infections; diarrhea; myeloid, renal and liver toxicity) associated with immunosuppressive therapy.
Prevalence of overlap syndromes and differential diagnoses | At baseline assessment and through study completion (up to 10 years)
  Reporting the prevalence of overlap syndromes and/or differential diagnoses with other primary or acquired cardias diseases other than myocarditis, including: arrhythmogenic cardiomyopathy (right, left, biventricular), dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy, noncompaction cardiomyopathy, toxic cardiomyopathy, ischemic cardiomyopathy; other genetic or acquired human diseases.
Comparison between histology abnormalities and arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Reporting the prevalence of any histological abnormality (normal vs. abnormal findings at either immunohistochemical, molecular, or ultrastructural analysis at EMB) in patients with arrhythmic vs. nonarrhythmic presentations of myocarditis.
Comparison between genetic test results and myocarditis features | At baseline assessment and through study completion (up to 10 years)
  Description, in genotyped patients, of any association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between genetic test results and myocarditis features (clinical presentation, associated diseases, findings at baseline workup, prognosis, and response to treatment).
Corrrelation between troponin abnormalities and follow-up occurrence of malignant ventricular arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between troponin abnormalities (ng/l) and occurrence of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy).
Corrrelation between troponin abnormalities and follow-up occurrence of heart failure | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between troponin abnormalities (ng/l) and occurrence of heart failure (= hospitalization for acute heart failure, heart transplantation, left ventricular ejection fraction below 35%).
Corrrelation between NTproBNP abnormalities and follow-up occurrence of malignant ventricular arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between NTproBNP abnormalities (pg/ml) and occurrence of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy).
Corrrelation between NTproBNP abnormalities and follow-up occurrence of heart failure | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between NTproBNP abnormalities (pg/ml) and occurrence of heart failure (= hospitalization for acute heart failure, heart transplantation, left ventricular ejection fraction below 35%).
Corrrelation between C-reactive protein abnormalities and follow-up occurrence of malignant ventricular arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between C-reactive protein abnormalities (mg/l) and occurrence of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy).
Corrrelation between C-reactive protein abnormalities and follow-up occurrence of heart failure | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between C-reactive protein abnormalities (mg/l) and occurrence of heart failure (= hospitalization for acute heart failure, heart transplantation, left ventricular ejection fraction below 35%).
Corrrelation between histological abnormalities and follow-up occurrence of malignant ventricular arrhythmias | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between histological abnormalities (any abnormality including immunohistochemical, molecular, and ultrastructural findings) and occurrence of malignant ventricular arrhythmias (= VT, VF, appropriate ICD therapy).
Corrrelation between histological abnormalities and follow-up occurrence of heart failure | At baseline assessment and through study completion (up to 10 years)
  Reporting the association (in terms of sensitivity, specificity, positive predictive value, negative predictive value) between histological abnormalities (any abnormality including immunohistochemical, molecular, and ultrastructural findings) and occurrence of heart failure (= hospitalization for acute heart failure, heart transplantation, left ventricular ejection fraction below 35%).
Comparison of minor arrhythmic events in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of the occurrence of minor arrhythmic events (NSVT; PVC burden; supraventricular arrhythmias; bradyarrhythmias) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of left ventricular end-diastolic volume in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of left ventricular end-diastolic volume (LVEDVi, ml/m2) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of right ventricular end-diastolic volume in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of right ventricular end-diastolic volume (RVEDVi, ml/m2) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of left ventricular ejection fraction in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of left ventricular ejection fraction (LVEF, %) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of right ventricular ejection fraction in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of left ventricular ejection fraction (RVEF, %) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of biventricular global longitudinal strain in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of biventricular global longitudinal strain (GLS, %) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of left atrial volume in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of left atrial volume (LAVi, ml/m2) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of left ventricular diastolic dysfunction in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Evaluation of diastolic dysfunction (E/E' ratio) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of pericardial abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of pericardial abnormalities (presence of pericardial effusion) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of valvular abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of valvular abnormalities (presence of valvular disease) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of CMR abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of CMR abnormalities (classic and modern Lake Louise Criteria) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of DECT abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of DECT abnormalities (classic and modern Lake Louise Criteria) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of PET abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of PET abnormalities (abnormal FDG or ammonia uptake) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of electroanatomical mapping abnormalities in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of electroanatomical mapping abnormalities (low-voltage areas) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of symptoms in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Prevalence of symptoms in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of exercise tolerance in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in exercise tolerance (New York Heart Association class) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of troponin in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in troponin values (ng/l) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of NTproBNP in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in NTproBNP values (pg/ml) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of C-reactive protein in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in C-reactive protein values (mg/l) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of arrhythmia burden in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in arrhythmia burden (daily and montly incidence of arrhythmias) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of arrhythmia morphology in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in arrhythmia morphology (monomorphic vs. polymorphic) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of arrhythmia regularity in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in arrhythmia regularity (regular vs. irregular) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of arrhythmia tolerance in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Change in arrhythmia tolerance (presence vs. absence of syncope) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Evaluation of myocarditis healing time in patients undergoing different therapeutic strategies | At baseline assessment and through study completion (up to 10 years)
  Assessment of myocarditis healing time (months) in patient groups differing for:
  1-General cardiac treatment. 2-Specific aetiology-driven treatment. 3-Cardiac device implant. 4-Arrhythmia ablation.
Comparison of the incidence of minor arrhythmic events in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of the occurrence of minor arrhythmic events (NSVT; PVC burden; supraventricular arrhythmias; bradyarrhythmias) in different patient groups:
  A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of left ventricular ejection fraction in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of left ventricular ejection fraction (LVEF, %) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of CMR abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of CMR abnormalities (Lake Louise criteria positivity) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of DECT abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of DECT abnormalities (delayed enhancement positivity) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of PET abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of PET abnormalities (abnormal FDG or ammonia uptake) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of electroanatomical abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of electroanatomical mapping abnormalities (low-voltage areas/abnormal electrograms) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of troponin abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of troponin abnormalities (ng/l) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of NTproBNP abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of NTproBNP abnormalities (pg/ml) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of C-reactive protein abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of C-reactive protein abnormalities (mg/l) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of autoantibodies abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of autoantibodies (U/l) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of genetic test abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of genetic test abnormalities (mutations) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of histological abnormalities in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of histological abnormalities (presence/absence of abnormal findings at either immunohistochemical, molecular, or ultrastructural analyses) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of exercise tolerance in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of exercise tolerance (New York heart Association class) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups. C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of arrhythmia burden in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of arrhythmia burden (daily and monthly incidence of arrhythmias) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of arrhythmia morphology in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of 12-lead arrhythmia morphology (QRS axis) and their modification in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of arrhythmia regularity in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of arrhythmia regularity (cycle length variability) and their modification in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.
Comparison of myocarditis healing time in different patient subgroups | At baseline assessment and through study completion (up to 10 years)
  Evaluation of myocarditis healing time (months) in different patient groups: A. Arrhythmic myocarditis subgroups (1-4). B. Non-arrhythmic myocarditis subgroups (i.e.: fulminant, acute coronary syndrome-like, pericarditis-like, heart failure, nonischaemic dilated /hypokinetic cardiomyopathies of unknown aetiology…). C.Infectious vs. autoimmune vs. toxic myocarditis. D.Myocarditis treated by aetiology-based treatment vs. isolated cardiac medical treatment. E.Myocarditis at different disease stages: acute, hyperacute, fulminant, chronic active, post-inflammatory, or active vs. previous vs. non-myocarditis. F. Myocarditis presenting as organ-specific diseases vs. in the context of a genetic disorder or systemic disease. G.Myocarditis vs. peri-myocarditis/myo-pericarditis. H.Other subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Della Bella, MD, Study Chair — San Raffaele Scientific Institute, Milan, Italy
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests will be evaluated case by case by the PI.

REFERENCES:
- [Result] Ammirati E, Cipriani M, Moro C, Raineri C, Pini D, Sormani P, Mantovani R, Varrenti M, Pedrotti P, Conca C, Mafrici A, Grosu A, Briguglia D, Guglielmetto S, Perego GB, Colombo S, Caico SI, Giannattasio C, Maestroni A, Carubelli V, Metra M, Lombardi C, Campodonico J, Agostoni P, Peretto G, Scelsi L, Turco A, Di Tano G, Campana C, Belloni A, Morandi F, Mortara A, Ciro A, Senni M, Gavazzi A, Frigerio M, Oliva F, Camici PG; Registro Lombardo delle Miocarditi. Clinical Presentation and Outcome in a Contemporary Cohort of Patients With Acute Myocarditis: Multicenter Lombardy Registry. Circulation. 2018 Sep 11;138(11):1088-1099. doi: 10.1161/CIRCULATIONAHA.118.035319. PMID 29764898
- [Result] De Luca G, Campochiaro C, Franchini S, Sartorelli S, Candela C, Peretto G, Sala S, Dagna L. Unexpected acute lymphocytic virus-negative myocarditis in a patient with limited cutaneous systemic sclerosis: a case report. Scand J Rheumatol. 2019 Mar;48(2):166-167. doi: 10.1080/03009742.2018.1493744. Epub 2018 Sep 30. No abstract available. PMID 30269630
- [Result] Peretto G, Sala S, Rizzo S, De Luca G, Campochiaro C, Sartorelli S, Benedetti G, Palmisano A, Esposito A, Tresoldi M, Thiene G, Basso C, Della Bella P. Arrhythmias in myocarditis: State of the art. Heart Rhythm. 2019 May;16(5):793-801. doi: 10.1016/j.hrthm.2018.11.024. Epub 2018 Nov 24. PMID 30476544
- [Result] Peretto G, Sala S, De Luca G, Campochiaro C, Sartorelli S, Cappelletti AM, Rizzo S, Palmisano A, Esposito A, Margonato A, Tresoldi M, Thiene G, Basso C, Dagna L, Della Bella P. Impact of systemic immune-mediated diseases on clinical features and prognosis of patients with biopsy-proved myocarditis. Int J Cardiol. 2019 Apr 1;280:110-116. doi: 10.1016/j.ijcard.2018.11.104. Epub 2018 Nov 22. PMID 30522885
- [Result] Sartorelli S, De Luca G, Campochiaro C, Peretto G, Sala S, Esposito A, Busnardo E, Basso C, Thiene G, Dagna L. Successful use of sirolimus in a patient with cardiac microangiopathy in primary antiphospholipid syndrome. Scand J Rheumatol. 2019 Nov;48(6):515-516. doi: 10.1080/03009742.2019.1574022. Epub 2019 Feb 22. No abstract available. PMID 30794015
- [Result] Gatti M, Palmisano A, Faletti R, Benedetti G, Bergamasco L, Bioletto F, Peretto G, Sala S, De Cobelli F, Fonio P, Esposito A. Two-dimensional and three-dimensional cardiac magnetic resonance feature-tracking myocardial strain analysis in acute myocarditis patients with preserved ejection fraction. Int J Cardiovasc Imaging. 2019 Jun;35(6):1101-1109. doi: 10.1007/s10554-019-01588-8. Epub 2019 Mar 30. PMID 30929101
- [Result] De Luca G, Campochiaro C, Sartorelli S, Peretto G, Sala S, Palmisano A, Esposito A, Candela C, Basso C, Rizzo S, Thiene G, Della Bella P, Dagna L. Efficacy and safety of mycophenolate mofetil in patients with virus-negative lymphocytic myocarditis: A prospective cohort study. J Autoimmun. 2020 Jan;106:102330. doi: 10.1016/j.jaut.2019.102330. Epub 2019 Sep 3. PMID 31488318
- [Result] Peretto G, Basso C, Bella PD, Sala S. Thyroid dysfunction in adult patients with biopsy-proved myocarditis: Screening and characterization. Eur J Intern Med. 2020 Jan;71:98-100. doi: 10.1016/j.ejim.2019.11.008. Epub 2019 Nov 14. No abstract available. PMID 31733987
- [Result] Campochiaro C, De Luca G, Tomelleri A, Sartorelli S, Peretto G, Sala S, Palmisano A, Esposito A, Cavalli G, Dagna L. Tocilizumab for the Treatment of Myocardial Inflammation Shown by Cardiac Magnetic Resonance: Report of Two Cases and Rationale for Its Therapeutic Use. J Clin Rheumatol. 2021 Dec 1;27(8S):S476-S479. doi: 10.1097/RHU.0000000000001194. No abstract available. PMID 31790000
- [Result] De Luca G, Campochiaro C, De Santis M, Sartorelli S, Peretto G, Sala S, Canestrari G, De Lorenzis E, Basso C, Rizzo S, Thiene G, Palmisano A, Esposito A, Selmi C, Gremese E, Della Bella P, Dagna L, Bosello SL. Systemic sclerosis myocarditis has unique clinical, histological and prognostic features: a comparative histological analysis. Rheumatology (Oxford). 2020 Sep 1;59(9):2523-2533. doi: 10.1093/rheumatology/kez658. PMID 31990340
- [Result] Peretto G, Sala S, Basso C, Della Bella P. Programmed ventricular stimulation in patients with active vs previous arrhythmic myocarditis. J Cardiovasc Electrophysiol. 2020 Mar;31(3):692-701. doi: 10.1111/jce.14374. Epub 2020 Feb 3. PMID 31999020
- [Result] Peretto G, Sala S, Della Bella P. [Diagnostic and therapeutic approach to myocarditis patients presenting with arrhythmias]. G Ital Cardiol (Rome). 2020 Mar;21(3):187-194. doi: 10.1714/3306.32767. Italian. PMID 32100731
- [Result] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Result] Palmisano A, Benedetti G, Faletti R, Rancoita PMV, Gatti M, Peretto G, Sala S, Boccia E, Francone M, Galea N, Basso C, Del Maschio A, De Cobelli F, Esposito A. Early T1 Myocardial MRI Mapping: Value in Detecting Myocardial Hyperemia in Acute Myocarditis. Radiology. 2020 May;295(2):316-325. doi: 10.1148/radiol.2020191623. Epub 2020 Mar 10. PMID 32154772
- [Result] Sala S, Peretto G, Gramegna M, Palmisano A, Villatore A, Vignale D, De Cobelli F, Tresoldi M, Cappelletti AM, Basso C, Godino C, Esposito A. Acute myocarditis presenting as a reverse Tako-Tsubo syndrome in a patient with SARS-CoV-2 respiratory infection. Eur Heart J. 2020 May 14;41(19):1861-1862. doi: 10.1093/eurheartj/ehaa286. No abstract available. PMID 32267502
- [Result] Peretto G, Sala S, Lazzeroni D, Palmisano A, Gigli L, Esposito A, De Cobelli F, Camici PG, Mazzone P, Basso C, Della Bella P. Septal Late Gadolinium Enhancement and Arrhythmic Risk in Genetic and Acquired Non-Ischaemic Cardiomyopathies. Heart Lung Circ. 2020 Sep;29(9):1356-1365. doi: 10.1016/j.hlc.2019.08.018. Epub 2019 Nov 15. PMID 32299760
- [Result] Palmisano A, Vignale D, Peretto G, Busnardo E, Calcagno C, Campochiaro C, De Luca G, Sala S, Ferro P, Basso C, Del Maschio A, De Cobelli F, Esposito A. Hybrid FDG-PET/MR or FDG-PET/CT to Detect Disease Activity in Patients With Persisting Arrhythmias After Myocarditis. JACC Cardiovasc Imaging. 2021 Jan;14(1):288-292. doi: 10.1016/j.jcmg.2020.03.009. Epub 2020 Apr 15. No abstract available. PMID 32305473
- [Result] Peretto G, Casella M, Merlo M, Benedetti S, Rizzo S, Cappelletto C, Di Resta C, Compagnucci P, De Gaspari M, Dello Russo A, Casari G, Basso C, Sala S, Sinagra G, Della Bella P, Cooper LT Jr. Inflammation on Endomyocardial Biopsy Predicts Risk of MACE in Undefined Left Ventricular Arrhythmogenic Cardiomyopathy. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 1):951-961. doi: 10.1016/j.jacep.2022.10.032. Epub 2023 Jan 18. PMID 36752457
- [Result] Peretto G, Maranta F, Cianfanelli L, Sala S, Cianflone D. Outcomes of inflammatory cardiomyopathy following cardiac rehabilitation. J Cardiovasc Med (Hagerstown). 2023 Jan 1;24(1):59-61. doi: 10.2459/JCM.0000000000001388. No abstract available. PMID 36574301
- [Result] Palmisano A, Vignale D, Bruno E, Peretto G, De Luca G, Campochiaro C, Tomelleri A, Agricola E, Montorfano M, Esposito A. Cardiac magnetic resonance findings in acute and post-acute COVID-19 patients with suspected myocarditis. J Clin Ultrasound. 2023 May;51(4):613-621. doi: 10.1002/jcu.23416. Epub 2022 Dec 21. PMID 36544331
- [Result] Peretto G, Gulletta S, Slavich M, Campochiaro C, Vignale D, De Luca G, Palmisano A, Villatore A, Rizzo S, Cavalli G, De Gaspari M, Busnardo E, Gianolli L, Dagna L, Basso C, Esposito A, Sala S, Della Bella P, Mazzone P. Exercise Stress Test Late after Arrhythmic versus Nonarrhythmic Presentation of Myocarditis. J Pers Med. 2022 Oct 12;12(10):1702. doi: 10.3390/jpm12101702. PMID 36294841
- [Result] Peretto G, Busnardo E, Ferro P, Palmisano A, Vignale D, Esposito A, De Luca G, Campochiaro C, Sartorelli S, De Gaspari M, Rizzo S, Dagna L, Basso C, Gianolli L, Della Bella P, Sala S. Clinical Applications of FDG-PET Scan in Arrhythmic Myocarditis. JACC Cardiovasc Imaging. 2022 Oct;15(10):1771-1780. doi: 10.1016/j.jcmg.2022.02.029. Epub 2022 May 11. PMID 36202457
- [Result] Ammirati E, Raimondi F, Piriou N, Sardo Infirri L, Mohiddin SA, Mazzanti A, Shenoy C, Cavallari UA, Imazio M, Aquaro GD, Olivotto I, Pedrotti P, Sekhri N, Van de Heyning CM, Broeckx G, Peretto G, Guttmann O, Dellegrottaglie S, Scatteia A, Gentile P, Merlo M, Goldberg RI, Reyentovich A, Sciamanna C, Klaassen S, Poller W, Trankle CR, Abbate A, Keren A, Horowitz-Cederboim S, Cadrin-Tourigny J, Tadros R, Annoni GA, Bonoldi E, Toquet C, Marteau L, Probst V, Trochu JN, Kissopoulou A, Grosu A, Kukavica D, Trancuccio A, Gil C, Tini G, Pedrazzini M, Torchio M, Sinagra G, Gimeno JR, Bernasconi D, Valsecchi MG, Klingel K, Adler ED, Camici PG, Cooper LT Jr. Acute Myocarditis Associated With Desmosomal Gene Variants. JACC Heart Fail. 2022 Oct;10(10):714-727. doi: 10.1016/j.jchf.2022.06.013. Epub 2022 Sep 7. PMID 36175056
- [Result] Ramirez GA, Batani V, Moroni L, De Luca G, Pizzetti G, Sala S, Peretto G, Campochiaro C, Della-Torre E, Bozzolo EP, Dagna L. Cardiac Safety of mRNA-Based Vaccines in Patients with Systemic Lupus Erythematosus and Lupus-like Disorders with a History of Myocarditis. Pathogens. 2022 Sep 1;11(9):1001. doi: 10.3390/pathogens11091001. PMID 36145434
- [Result] Peretto G, Merlo M, Gentile P, Porcari A, Palmisano A, Vignale D, Sormani P, Rizzo S, De Gaspari M, Basso C, Bella PD, Sala S, Ammirati E, Sinagra G, Esposito A, Pedrotti P. Cardiac magnetic resonance abnormalities in patients with acute myocarditis proven by septal endomyocardial biopsy. Clin Res Cardiol. 2023 Mar;112(3):392-400. doi: 10.1007/s00392-022-02103-1. Epub 2022 Sep 16. PMID 36112234
- [Result] Nowatzke J, Guedeney P, Palaskas N, Lehmann L, Ederhy S, Zhu H, Cautela J, Francis S, Courand PY, Deswal A, Ewer SM, Aras M, Arangalage D, Ghafourian K, Fenioux C, Finke D, Peretto G, Zaha V, Itzhaki Ben Zadok O, Tajiri K, Akhter N, Levenson J, Baldassarre L, Power J, Huang S, Collet JP, Moslehi J, Salem JE; International ICI-myocarditis registry contributors. Coronary artery disease and revascularization associated with immune checkpoint blocker myocarditis: Report from an international registry. Eur J Cancer. 2022 Dec;177:197-205. doi: 10.1016/j.ejca.2022.07.018. Epub 2022 Aug 24. PMID 36030143
- [Result] Villatore A, Sala S, Stella S, Vignale D, Busnardo E, Esposito A, Basso C, Della Bella P, Mazzone P, Peretto G. Autoimmune Myocarditis and Arrhythmogenic Mitral Valve Prolapse: An Unexpected Overlap Syndrome. J Cardiovasc Dev Dis. 2021 Nov 6;8(11):151. doi: 10.3390/jcdd8110151. PMID 34821704
- [Result] Campochiaro C, Tomelleri A, Farina N, Cavalli G, De Luca G, Palmisano A, Peretto G, Esposito A, Rizzo S, Basso C, Matucci-Cerinic M, Dagna L. Myocarditis as a manifestation of Erdheim-Chester Disease: successful use of anti- IL1 and BRAF inhibitor combination therapy. Scand J Rheumatol. 2022 May;51(3):243-245. doi: 10.1080/03009742.2021.1992846. Epub 2021 Nov 17. No abstract available. PMID 34788207
- [Result] Peretto G, Mazzone P, Paglino G, Marzi A, Tsitsinakis G, Rizzo S, Basso C, Della Bella P, Sala S. Continuous Electrical Monitoring in Patients with Arrhythmic Myocarditis: Insights from a Referral Center. J Clin Med. 2021 Nov 1;10(21):5142. doi: 10.3390/jcm10215142. PMID 34768662
- [Result] Campochiaro C, Farina N, Tomelleri A, Ferrara R, Lazzari C, De Luca G, Bulotta A, Signorelli D, Palmisano A, Vignale D, Peretto G, Sala S, Esposito A, Garassino M, Gregorc V, Dagna L. Tocilizumab for the treatment of immune-related adverse events: a systematic literature review and a multicentre case series. Eur J Intern Med. 2021 Nov;93:87-94. doi: 10.1016/j.ejim.2021.07.016. Epub 2021 Aug 12. PMID 34391591
- [Result] Gentile P, Merlo M, Peretto G, Ammirati E, Sala S, Della Bella P, Aquaro GD, Imazio M, Potena L, Campodonico J, Foa A, Raafs A, Hazebroek M, Brambatti M, Cercek AC, Nucifora G, Shrivastava S, Huang F, Schmidt M, Muser D, Van de Heyning CM, Van Craenenbroeck E, Aoki T, Sugimura K, Shimokawa H, Cannata A, Artico J, Porcari A, Colopi M, Perkan A, Bussani R, Barbati G, Garascia A, Cipriani M, Agostoni P, Pereira N, Heymans S, Adler ED, Camici PG, Frigerio M, Sinagra G. Post-discharge arrhythmic risk stratification of patients with acute myocarditis and life-threatening ventricular tachyarrhythmias. Eur J Heart Fail. 2021 Dec;23(12):2045-2054. doi: 10.1002/ejhf.2288. Epub 2021 Jul 21. PMID 34196079
- [Result] Peretto G, Cappelletti AM, Spoladore R, Slavich M, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Margonato A, Basso C, Della Bella P, Sala S. Right ventricular endomyocardial biopsy in patients with cardiac magnetic resonance showing left ventricular myocarditis. J Cardiovasc Med (Hagerstown). 2021 Jul 1;22(7):560-566. doi: 10.2459/JCM.0000000000001162. PMID 34076604
- [Result] Peretto G, Villatore A, Rizzo S, Esposito A, De Luca G, Palmisano A, Vignale D, Cappelletti AM, Tresoldi M, Campochiaro C, Sartorelli S, Ripa M, De Gaspari M, Busnardo E, Ferro P, Calabro MG, Fominskiy E, Monaco F, Cavalli G, Gianolli L, De Cobelli F, Margonato A, Dagna L, Scandroglio M, Camici PG, Mazzone P, Della Bella P, Basso C, Sala S. The Spectrum of COVID-19-Associated Myocarditis: A Patient-Tailored Multidisciplinary Approach. J Clin Med. 2021 May 4;10(9):1974. doi: 10.3390/jcm10091974. PMID 34064463
- [Result] Peretto G, Sala S, Camaschella C. Iron deficiency in chronic myocarditis: Assessment and prognostic significance. Eur J Intern Med. 2021 Jul;89:129-131. doi: 10.1016/j.ejim.2021.03.037. Epub 2021 Apr 21. No abstract available. PMID 33893018
- [Result] Peretto G, Barzaghi F, Cicalese MP, Di Resta C, Slavich M, Benedetti S, Giangiobbe S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Gulletta S, Basso C, Casari G, Aiuti A, Della Bella P, Sala S. Immunosuppressive therapy in childhood-onset arrhythmogenic inflammatory cardiomyopathy. Pacing Clin Electrophysiol. 2021 Mar;44(3):552-556. doi: 10.1111/pace.14153. Epub 2021 Jan 18. PMID 33372694
- [Result] Cenciarelli S, Calbi V, Barzaghi F, Bernardo ME, Oltolini C, Migliavacca M, Gallo V, Tucci F, Fraschetta F, Albertazzi E, Fratini ES, Consiglieri G, Giannelli S, Dionisio F, Sartirana C, Racca S, Camesasca C, Peretto G, Daverio R, Esposito A, De Cobelli F, Silvani P, Rabusin M, Cara A, Trabattoni D, Dispinseri S, Scarlatti G, Piemonti L, Lampasona V, Cicalese MP, Aiuti A, Ferrua F. Mild SARS-CoV-2 Infection After Gene Therapy in a Child With Wiskott-Aldrich Syndrome: A Case Report. Front Immunol. 2020 Nov 24;11:603428. doi: 10.3389/fimmu.2020.603428. eCollection 2020. PMID 33329599
- [Result] Peretto G, Sala S, De Luca G, Marcolongo R, Campochiaro C, Sartorelli S, Tresoldi M, Foppoli L, Palmisano A, Esposito A, De Cobelli F, Rizzo S, Thiene G, Basso C, Dagna L, Caforio ALP, Della Bella P. Immunosuppressive Therapy and Risk Stratification of Patients With Myocarditis Presenting With Ventricular Arrhythmias. JACC Clin Electrophysiol. 2020 Oct;6(10):1221-1234. doi: 10.1016/j.jacep.2020.05.013. Epub 2020 Jun 24. PMID 33092747
- [Result] Peretto G, Sala S, Basso C, Rizzo S, Radinovic A, Frontera A, Limite LR, Paglino G, Bisceglia C, De Luca G, Campochiaro C, Sartorelli S, Palmisano A, Esposito A, Busnardo E, Villatore A, Baratto F, Cireddu M, Marzi A, D'Angelo G, Gulletta S, Vergara P, De Cobelli F, Dagna L, Mazzone P, Della Bella P. Inflammation as a Predictor of Recurrent Ventricular Tachycardia After Ablation in Patients With Myocarditis. J Am Coll Cardiol. 2020 Oct 6;76(14):1644-1656. doi: 10.1016/j.jacc.2020.08.012. PMID 33004129
- [Result] Peretto G, De Luca G, Campochiaro C, Palmisano A, Busnardo E, Sartorelli S, Barzaghi F, Cicalese MP, Esposito A, Sala S. Telemedicine in myocarditis: Evolution of a mutidisciplinary "disease unit" at the time of COVID-19 pandemic. Am Heart J. 2020 Nov;229:121-126. doi: 10.1016/j.ahj.2020.07.015. Epub 2020 Aug 12. PMID 32957030
- [Result] Peretto G, Sala S, Della Bella P, Basso C, Cooper LT Jr. Reply: Genetic Basis for Acute Myocarditis Presenting With Ventricular Arrhythmias? J Am Coll Cardiol. 2020 Jul 7;76(1):126-128. doi: 10.1016/j.jacc.2020.05.014. No abstract available. PMID 32616153

DOCUMENTS (1):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04521790/Prot_000.pdf